CLINICAL TRIAL: NCT03129126
Title: A Multicenter, Dose-Ranging Trial Evaluating the Safety, Tolerability and Efficacy of LP-10 in Subjects With Refractory Moderate to Severe Hemorrhagic Cystitis
Brief Title: The Safety, Tolerability and Efficacy of LP-10 in Subjects With Refractory Moderate to Severe Hemorrhagic Cystitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lipella Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: Safety and Efficacy of LP-10
Record Dates: First submitted 2017-04-17; First posted 2017-04-26 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-03

CONDITIONS: Hemorrhagic Cystitis
MeSH Terms: conditions — Cystitis, Hemorrhagic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LP-10 2mg (Experimental): LP-10 (intravesical tacrolimus), 2mg reconstituted in sterile water for injection, intravesical instillations, up to two instillations, instillations will occur greater than 3 days but less than 7 days apart as needed.
  Interventions: Drug: LP-10
- LP-10 4mg (Experimental): LP-10 (intravesical tacrolimus), 4mg reconstituted in sterile water for injection, intravesical instillations, up to two instillations, instillations will occur greater than 3 days but less than 7 days apart as needed.
  Interventions: Drug: LP-10
- LP-10 8mg (Experimental): LP-10 (intravesical tacrolimus), 8mg reconstituted in sterile water for injection, intravesical instillations, up to two instillations, instillations will occur greater than 3 days but less than 7 days apart as needed.
  Interventions: Drug: LP-10

INTERVENTIONS:
Drug: LP-10 — Intravesical tacrolimus

SUMMARY:
The purpose of this study is to assess the safety and tolerability of three doses of LP-10 (intravesical tacrolimus). Twelve subjects meeting the inclusion and exclusion criteria will be enrolled and treated in a prospective and multi-center trial with LP-10. The proposed trial will recruit 12 subjects in a dose-escalation trial where 4 subjects will be allocated into each one of three groups.

DETAILED DESCRIPTION:
This is a multi-center, dose-ranging study including male and female subjects with refractory moderate to severe hemorrhagic cystitis as determined by a physician. A total of up to 12 subjects are anticipated and will be enrolled in study sites in the United States. Enrollment is expected to be completed within one year of initiating the study. The proposed trial will recruit 12 subjects in a dose-escalation trial where 4 subjects will be allocated into each one of three groups.

ELIGIBILITY:
Inclusion Criteria:

Males and females, at least 18 years

* History of sterile moderate to severe HC (Grade 2-4) for at least 3 months documented in the medical record with at least 1 episode of macroscopic hematuria with or without clot
* Previous use of medications and/or treatment(s) for HC without success
* Patients of child-bearing capability agree to use a reliable form of birth control (condoms and/or oral contraceptives) during the course of instillation therapy and for 1 week thereafter
* Willing and capable of understanding and complying with all requirements of the protocol, including proper completion of the 3 day Hemorrhagic Cystitis Diary (HC Diary) and self-administered questionnaires

Exclusion Criteria:

* History of interstitial cystitis/painful bladder syndrome
* HC due to infection (bacterial, viral or fungal)
* Vesicoureteral reflux disease based on cystogram within past 12 months
* Subject is currently or has previously participated in another therapeutic or device study within 3 months of screening and has not returned to baseline
* Pregnant or lactating
* History of bleeding diathesis or active bleeding peptic ulcer disease
* Life expectancy less than 12 months
* PSA > 10.0 ng/dl (measured within the last 3 months)
* Known allergy to liposomes and/or egg yolk and/or tacrolimus
* Urinary retention requiring daily catheterization
* Previous augmentation cystoplasty
* Subjects currently taking prescribed treatment for HC will be able to continue the treatment throughout the course of the study. If the patient cannot be maintained on a stable dose of the medication(s) throughout the treatment and follow-up period they will be excluded
* Subject with history of intravesical treatment(s) within 1 week prior to Study Visit 1
* Sacral and/or pudendal nerve neuromodulation device (Interstim) within the last 6 months. Subjects would not be excluded if they had Interstim greater than 6 months ago and is on a stable setting.
* Evidence of renal impairment (creatinine > two times the upper limit of normal at Visit 1), hepatic impairment (AST or ALT > three times the upper limit of normal at Visit 1), clinically significant cardiovascular, respiratory, or psychiatric diseases per investigator's judgment
* Post-void residual (PVR) urine volume of > 150 mL at screening
* The presence of any clinically significant systemic disease or condition that in the opinion of the investigator would make the patient unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Patient Reported Mean episodes of visible blood | At every patient visit, up to 2 weeks following initial treatment
  Pre-post changes in mean episodes of visible blood in urine (or blood clots) on 3-day bladder diaries at baseline and primary endpoint

SECONDARY OUTCOMES:
Urine Dipstick Mean episodes of Visible Blood | At every patient visit, up to 2 weeks following initial treatment
  Mean episodes of visible blood in urine (or blood clots) and urine dipstick for quantitative grading of microscopic hematuria on bladder diaries
Mean urine hemoglobin concentration | At every patient visit, up to 2 weeks following initial treatment
  Mean urine hemoglobin concentration
Urine analysis with microscopy | At every patient visit, up to 2 weeks following initial treatment
  Urine analysis with microscopy including red blood cells per high power field test
Whole blood Add to dictionary levels | At every patient visit, up to 2 weeks following initial treatment
  Whole blood tacrolimus levels
Blood chemistry and liver function test | At every patient visit, up to 2 weeks following initial treatment
  Blood chemistry and liver function test
Patient Reported Global Response Assessment Survey Score | At every patient visit, up to 2 weeks following initial treatment
  Changes in Global Response Assessment (GRA)
Patient Reported Urinary frequency | At every patient visit, up to 2 weeks following initial treatment
  Changes in urinary frequency and incontinence measured on diaries
Bladder Cystoscopy | At initial treatment and on final patient visit, up to 2 weeks following initial treatment
  Cystoscopic changes in bladder
Patient Reported Health Related Quality of Life Survey Score | At every patient visit, up to 2 weeks following initial treatment
  Changes in Health Related Quality of Life (HRQOL) scores
Post void residual urine volume | At every patient visit, up to 2 weeks following initial treatment
  Post void residual urine volume
Patient Reported Pain and Urgency | At every patient visit, up to 2 weeks following initial treatment
  Change in pain and urgency 10 cm visual analog scales (VAS)
Incidence of Treatment-Emergent Adverse Events | At every patient visit, up to 2 weeks following initial treatment
  Safety data will be collected by ongoing monitoring of adverse events, during the entire duration of the study, including need for blood transfusion, bladder irrigation, emergency room visit, hospitalization, urinary catheterization, and/or surgery in addition to patient reporting of changes in urinary frequency, hematuria/ clots, incontinence, spasm or discomfort.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Arizona, Tucson, Arizona
  - University of California San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Michigan Institute of Urology, Troy, Michigan
  - Premier Medical Group, Poughkeepsie, New York
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny Health Network Research Institute, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided